CLINICAL TRIAL: NCT04120233
Title: A Phase 1a, Double-Blind, Randomized, Placebo-Controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetic Profile of MW151 Administered Orally to Healthy Volunteers
Brief Title: MW151-101: First-in-human Study of MW151
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Linda Van Eldik (Other)
Collaborators: Duke Clinical Research Institute (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Linda Van Eldik, Director, Sanders-Brown Center on Aging, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: Pro00103072, IND143222; R01AG061898 (NIH)
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Drug Toxicity
Keywords: cognitive disorder; pharmacokinetics; MW151; MW01-2-151SRM; PK; dose escalation
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Cognitive Dysfunction | interventions — 2-(4-(4-methyl-6-phenylpyridazin-3-yl)piperazin-1-yl)pyrimidine

STUDY DESIGN:
Intervention Model Description: Dose-escalation study.
Who Masked: Outcomes Assessor
Masking Description: Data from cohorts will be reviewed in a blinded manner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo
- Dose 1 (Experimental): Participants will receive 10 mg of MW151.
  Interventions: Drug: MW151, 10mg
- Dose 2 (Experimental): Participants will receive 20mg of MW151.
  Interventions: Drug: MW151, 20mg
- Dose 3 (Experimental): Participants will receive 40mg of MW151.
  Interventions: Drug: MW151, 40mg
- Dose 4 (Experimental): Participants will receive 80mg of MW151.
  Interventions: Drug: MW151, 80mg
- Dose 5 (Experimental): Participants will receive 160mg of MW151.
  Interventions: Drug: MW151, 160mg

INTERVENTIONS:
Drug: Placebo — Matched placebo administered orally
  Arms: Placebo
Drug: MW151, 10mg — 10 mg MW151, 1 x 10mg capsule administered orally
  Arms: Dose 1
Drug: MW151, 20mg — 20 mg MW151, 1 x 20mg capsule administered orally
  Arms: Dose 2
Drug: MW151, 40mg — 40 mg MW151, 2 x 20mg capsule administered orally
  Arms: Dose 3
Drug: MW151, 80mg — 80 mg MW151, 1 x 80mg capsule administered orally
  Arms: Dose 4
Drug: MW151, 160mg — 160 mg MW151, 2 x 80mg capsule administered orally
  Arms: Dose 5

SUMMARY:
MW01-2-151SRM (=MW151), a small molecule, is being developed for the treatment of cognitive disorders. The development program is based on nonclinical evidence that MW151 improves neurocognitive outcomes in animal models of radiation-induced cognitive impairment, Alzheimer's disease, and other central nervous system (CNS) disorders.

The present study will provide safety and pharmacokinetic (PK) information on single ascending doses to support decisions for continued clinical development.

DETAILED DESCRIPTION:
The primary objective of this trial is to assess the safety and tolerability of single ascending doses of MW151 when administered orally to healthy adults.

Subjects will be screened prior to inpatient admission. Subjects will be admitted to the inpatient clinic on the day prior to dosing (Day -1) and will remain in the unit until discharge on Day 3. A follow-up visit will be done on Day 7. A single dose of study drug or placebo will be administered on Day 1. Healthy adult female subjects will be randomly assigned to one of 5 dose cohorts (8 subjects each). Each subject will receive a single dose of MW151 (10-160mg) or placebo under fasted conditions.

Following a review of safety and tolerability data for the first 24 hours of dosing in each cohort (including reported adverse events (AEs), physical examination findings, clinical laboratory results, vital signs, and electrocardiograms (ECGs), the remaining 6 subjects will be randomized in a 5:1 ratio. Dosing of the remaining subjects in a cohort may proceed after review of sentinel subject safety data collected during the first 24 hours of dosing and determination that no stopping rules are met. The remaining subjects in each cohort will be dosed sequentially, not simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* In good health as determined by medical history, physical exam, laboratory examinations, ECG, and vital signs.
* Weight >50kg
* BMI <34 kg/m2.
* ECG without clinically significant pathologic abnormalities and with QTcF <450 ms -
* Systolic BP ≤ 150 mmHg and diastolic BP ≤ 90 mmHg at screening
* No suicidal ideation, as demonstrated by a score of "0" on the Columbia Suicide Severity Rating Scale (C-SSRS).
* Women who are neither pregnant (negative pregnancy test) nor nursing, and are either: surgically sterile, postmenopausal with last natural menses greater than 24 months, or premenopausal and agrees to use and acceptable form of birth control during the study and for 1 month after dosing.
* Adequate venous access for blood draws.

Exclusion Criteria:

* Any unstable chronic medical condition requiring interventional treatment that might increase the risk to the subject or confound interpretation of safety observations. Subjects who are considered stable and who have been receiving stable treatment for medical condition for > 3 months may be considered with approval of medical monitor.
* Evidence of active infection requiring antibiotic therapy within 14 days prior to dosing.
* Medical history of vasculitis or any autoimmune disease excluding seasonal allergic rhinitis and childhood history of atopic dermatitis.
* History of any treatment for cancer within the past 2 years, other than basal cell or squamous cell carcinoma of the skin.
* Seropositive for human immunodeficiency virus (HIV).
* History of acute/chronic hepatitis B or C and/or carriers of hepatitis B
* Clinically significant abnormalities in screening laboratory tests
* Over-the-counter and herbal medications are prohibited within 10 days prior to study dosing (with exception of calcium/vitamin D supplements and ocular medications at the discretion of the Investigator). Stable doses (> to 3 months of stable dose) of prescription medications are allowed with the approval of the medical monitor (birth control medications are allowed without medical monitor approval). Subjects should not be on non-steroidal anti-inflammatory drugs or immunosuppressive drugs within 10 days prior to dosing.
* Use of known CYP450 CYP1A2, CYP2D6 or CYP3A4 inhibitors or inducers within 14 days of dosing or planned use during the study.
* Use of an investigational drug, vaccine, device, or blood product within 3 months prior to dosing in this study.
* Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g. small bowel disease, Crohn's disease, celiac disease, or liver disease.)
* Psychiatric history of current or past psychosis, bi-polar disorder, clinical depression, or anxiety disorder requiring chronic medication within the past 5 years.
* History of substance abuse including alcohol within the past 5 years.
* Smoker.
* Current substance or drug dependence confirmed by positive urine drug screen at screening visit or Day -1 admission.
* Current alcohol abuse confirmed by positive breathalyzer at screening visit or Day -1 admission.
* History of serious head injury as determined by the site investigator or designee.
* Chronic kidney disease (defined as the presence of any degree of proteinuria on urine analysis and/or an eGFR of <60 ml/min using the MDRD formula).
* Any reason or opinion of the investigator that would prevent the subject from participation in the study.
* Inability to follow the instructions or an unwillingness to cooperate with study procedures.
* Has donated more than 500 mL of blood within the last month prior to dosing.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-09-16 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Van Eldik, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated on October 11, 2019 and last follow-up was completed on September 16,2021.
Pre-assignment Details: A total of 97 subjects were screened and 40 subjects were randomized.
Period: Overall Study
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
Started | 10 | 6 | 6 | 6 | 6 | 6
Completed | 10 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5 | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (9.4) | 37.9 (8.3) | 39.3 (8.2) | 34.5 (8.6) | 40.9 (6.4) | 35.2 (7.4) | 36.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 6 | 6 | 6 | 6 | 33
  Male | 1 | 6 | 0 | 0 | 0 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 0 | 1 | 0 | 7
  Not Hispanic or Latino | 7 | 6 | 3 | 6 | 5 | 6 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 1 | 2 | 2 | 5 | 17
  White | 5 | 3 | 4 | 3 | 2 | 1 | 18
  More than one race | 1 | 0 | 0 | 1 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 6 | 6 | 6 | 6 | 40
Height [Mean (Standard Deviation); unit: cm] | 163.3 (5.8) | 178.1 (8.2) | 158.0 (7.5) | 162.5 (1.9) | 169.3 (7.5) | 165.1 (4.3) | 165.9 (8.5)
Weight [Mean (Standard Deviation); unit: kg] | 74.8 (11.7) | 85.3 (15.2) | 70.5 (12.9) | 68.1 (7.6) | 79.6 (17.4) | 75.1 (10.2) | 75.5 (13.1)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (3.6) | 26.9 (3.8) | 28.3 (4.9) | 25.8 (2.6) | 27.5 (4.3) | 27.6 (4.0) | 27.4 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Drug-related Serious Adverse Events.
Description: Percentage of participants experiencing drug-related serious adverse events from the start of study drug administration up to 7-day follow-up.
Time Frame: Seven days
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Drug Concentration (Cmax)
Description: Peak serum concentration of MW151.
Time Frame: predose, 0.25h, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h and 36h post-dose
Population: The PK population included all subjects who were administered MW151 and had at least 1 quantifiable concentration of MW151 measurement.
  One subject in Cohort 4 withdrew prior to the 36h plasma sampling, so that sampling point was excluded from the PK dataset at that timepoint.
  PK parameters for MW151 cannot be analyzed in the placebo group, as they did not receive the study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6
ng/mL |  | 32.2 (14.6) | 132.0 (62.5) | 283.0 (244) | 361.0 (53.2) | 1190.0 (707.0)

3. Secondary Outcome: Time to Maximum Drug Concentration (Tmax)
Description: Time required to reach the maximum serum concentration of MW151.
Time Frame: predose, 0.25h, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h and 36h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6
hours |  | 1.8 (0.4) | 1.6 (0.7) | 1.5 (1.4) | 2.3 (1.4) | 2.0 (1.6)

4. Secondary Outcome: Overall Drug Exposure (AUC)
Description: Overall drug exposure (h*ng/mL) determined by calculating the area under the curve (AUC) from a plasma drug concentration-time curve.
Time Frame: predose, 0.25h, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h and 36h post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 6
h*ng/mL |  | 208.0 (91.8) | 741.0 (168.0) | 1250.0 (453.0) | 3120.0 (1290.0) | 7590.0 (1800.0)

5. Secondary Outcome: Drug Half-Life (T1/2)
Description: Time at which the concentration of MW151 is at half the maximum concentration.
Time Frame: predose, 0.25h, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h and 36h post-dose
Population: Placebo: PK parameters for MW151 cannot be analyzed, as they did not receive the study drug.
  Dose 2: Data from two participants were excluded for being nonacceptable, and were not analyzed.
  Dose 3, 4 and 5: Data from 5 participants in each group were nonacceptable, and were not analyzed.
  Non-acceptance data are defined as: R^2_adjusted <0.8 and terminal elimination phase time span <3 half-lives after Tmax.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
Number analyzed (Participants) | 0 | 6 | 4 | 1 | 1 | 1
hour |  | 8.2 (1.9) | 10.6 (1.4) | 8.8 (NA) — Only one participant did not have non-acceptance data. Since data from only one participant was analyzed the deviation cannot be calculated. | 10.4 (NA) — Only one participant did not have non-acceptance data. Since data from only one participant was analyzed the deviation cannot be calculated. | 10.6 (NA) — Only one participant did not have non-acceptance data. Since data from only one participant was analyzed the deviation cannot be calculated.

6. Secondary Outcome: Elimination Rate Constant (Kel)
Description: Fraction of MW151 eliminated per unit of time (mathematical determination).
Time Frame: predose, 0.25h, 0.5h, 1h, 2h, 4h, 8h, 12h, 24h and 36h post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
Number analyzed (Participants) | 0 | 6 | 4 | 1 | 1 | 1
1/h |  | 0.09 (0.02) | 0.07 (0.01) | 0.08 (NA) — Only one participant did not have non-acceptance data. Since data from only one participant was analyzed the deviation cannot be calculated. | 0.07 (NA) — Only one participant did not have non-acceptance data. Since data from only one participant was analyzed the deviation cannot be calculated. | 0.07 (NA) — Only one participant did not have non-acceptance data. Since data from only one participant was analyzed the deviation cannot be calculated.

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to 7-day follow-up
Arm/Group | Placebo | Dose 1 | Dose 2 | Dose 3 | Dose 4 | Dose 5
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/10 | 0/6 | 4/6 | 3/6 | 3/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Dose 1 (N=6) | Dose 2 (N=6) | Dose 3 (N=6) | Dose 4 (N=6) | Dose 5 (N=6)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 3 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04120233/Prot_SAP_ICF_000.pdf